CLINICAL TRIAL: NCT02069639
Title: Serum Thymus and Activation-regulated Chemokine (TARC) Level Monitoring May Predict Disease Relapse Detected by PET Scan After Reduced Intensity Allogeneic Stem Cell Transplantation in Hodgkin's Lymphoma Patients
Brief Title: TARC After alloSCT in Hodgkin's Lymphoma
Acronym: TARC
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Paolo Corradini, md, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: TARC
Record Dates: First submitted 2014-02-14; First posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Hodgkin's Lymphoma Patients Who Underwent an Allogeneic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- no treatment
  Interventions: Other: no treatment

INTERVENTIONS:
Other: no treatment

SUMMARY:
Relapsed and refractory Hodgkin's lymphoma (HL) patients may experience long-term survival after allogeneic transplant (alloSCT), but disease recurrence represents the main cause of treatment failure. PET (positron-emission tomography) -positive patients after alloSCT have a dismal outcome. Serum TARC (thymus and activation-regulated chemokine) is produced by Reed-Sternberg cells and may be a marker of disease. Our study was aimed at assessing whether TARC levels after alloSCT were correlated to disease status and whether TARC monitoring could increase the ability to predict relapse.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin's lymphoma patients who underwent an alloSCT at Fondazione IRCCS Istituto Nazionale dei Tumori and who were monitored by PET and TARC before and after alloSCT from 2009

Exclusion Criteria:

* Hodgkin's lymphoma patients who underwent an alloSCT who were not monitored by PET or/and TARC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 22 consecutive Hodgkin's lymphoma patients who underwent an alloSCT at Fondazione IRCCS Istituto Nazionale dei Tumori and who were monitored by PET and TARC before and after alloSCT.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Correlation between disease status and serum TARC level | One year after transplant
  Serum TARC level was measured before alloSCT in Hodgkin's lymphoma patients and after alloSCT. The median time interval after alloSCT was 47 days. PFS was estimated at one year based on TARC value.

SECONDARY OUTCOMES:
The correlation between TARC levels and PET results after alloSCT | Before alloSCT, monthly during the first 6 months after alloSCT and every 2 months until 2 years of follow-up, then at the time of clinical check-up (usually every 6 months)
  We selected TARC values done on the days of PET to assess a cut-off value of TARC that was correlated to a positive or negative PET

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy